Document Date: 03/22/2021

NCT# NCT04913363

# Consent of an Adult to Be in a Research Study

In this form "you" means a person 18 years of age or older who is being asked to volunteer to participate in this study.

| Participant's | Name | <b>!</b> |
|---------------|------|----------|

## What is the purpose of this form?

This form will provide you with information about this research study. You do not have to be in the study if you do not want to. You should have all your questions answered before you agree to be in this study.

Please read this form carefully. If you want to be in the study, you will need to sign this form. You will be given a copy of this form.

# Who is funding this study?

This study is funded by a grant from the iThriv Community Engaged Research, from the National Institute of Health (NIH).

## **Key Information About This Research Study**

This study aims to understand the impact of different outdoor activities on health and wellbeing in JABA service users. To this end, we will compare responses to a series of survey questions both before and after a short activity (walking, citizen science – a guided, interactive walk - and planting) as well as recording your movement using a wearable accelerometer. For two of these sessions, we will transport you via a Jaunt bus from the Mary Williams Senior Community Center to Wild Rock Nature Preserve. If you would like to make your own travel arrangements, this is no problem and can be discussed if you choose to sign up.

We will ask you to attend three separate sessions in which you will complete one of the three activities. You will complete a different activity in each session, after which you will be compensated with a \$10 supermarket voucher for each of the three sessions you complete. There are no benefits to you for completing this study.

All study sessions will follow strict COVID-19 safety protocols and we ask you comply with these, including face mask wearing at all times, clean hands between activities and social distance throughout.

UVA Study Tracking: HSR210100

Version Date: 03-22-21 Page Number: 1 of 7

| Principal Investigator: | Professor Jennifer Roe, Director, Center for Design and Health, |
|---|---|
| | School of Architecture, 418 Campbell Hall, PO Box 400122, |
| | University of Virginia, Charlottesville, VA 22904. |
| | Telephone: (434) 242 4567 |
| | Email: jjr4b@virginia.edu |

You are being asked to take part in a research study. You do not have to take part in this study. You should only agree to take part in this study after reading this consent form and discussing it with the study team. You may also discuss this with your family, friends, health care providers or others before you make a decision.

#### What problem is this study trying to solve?

This study is trying to find out if there is any benefit of outdoor activities on health and wellbeing of JABA service users. You are being asked to take part in this study because you are, or have been, a JABA service user.

#### Why would you want to take part in this study?

You will not be helped by being in this study, but the information gained by doing this study may help others in the future. This information may inform future JABA activities.

#### Why would you NOT want to take part in this study?

You might not want to take part in this study because, as with any outdoor activity in your local area, there are risks of falling or traffic accidents. However, we do not anticipate any greater risk to you than you would have on a normal walk in your local environment. We will attempt to highlight any specific risks on the testing day both verbally and by making chalk marks on the sidewalk.

#### What will I have to do if I take part in this study?

Full details of all the procedures are found later in this form. If you take part in this study you will be asked to complete a short survey consisting of demographic, mood, comfort and health questions. You will be asked to repeat these after completing one of three activities around the local area. During these activities, you will be wearing a sensor that will record movement. It is anticipated that each of the three sessions will last for a maximum of sixty minutes (including briefing, transport and the measures themselves).

UVA Study Tracking: HSR210100

Version Date: 03-22-21 Page Number: 2 of 7

## What will happen if you are in the study?

If you agree to participate, you will sign this consent form before any study related procedures take place.

You will complete three different activities, each on a separate day. One will be a walking session were you will walk a predetermined route around a local nature preserve. The second will be a citizen science walk, where a trained citizen scientist will talk you through points of interest in a local green space. The third activity will be a planting session where a master gardener will give you a tutorial in planting and tending to plants at the JABA center. These sessions will be roughly one week apart. We advise you wear comfortable clothes that you can be mildly active in, suitable for the weather conditions of the day.

You will compete questionnaires before and after each activity. These questionnaires ask about:

- Demographics (age, gender, etc.)
- Mood
- · Feelings of belonging and loneliness
- Physical activity and tiredness

These questionnaires will take about 10 minutes to complete.

During each activity, you will also be asked to wear an accelerometer which will measure your movement throughout the activity. The accelerometer is a wristband that you will leave on throughout the session.

# How long will this study take?

Your participation in this study will require 3 study visits over a three weeks. Each visit will last about 1 hour.

## What are the risks of being in this study?

As with any walk in your local area, there are risks of falling or traffic accidents. However, as this is an area you know, we do not anticipate any greater risk to you than you would have on a normal walk in your local environment. We will highlight any specific risks on the testing day both verbally and by making chalk marks on the sidewalk.

## Could you be helped by being in this study?

You will not benefit from being in this study. However, the information researchers get from this study may help others in the future.

UVA Study Tracking: HSR210100

Version Date: 03-22-21 Page Number: 3 of 7

#### What are your other choices if you do not join this study?

The only choice is not to be in this study. You are free to withdraw at any time.

## Will you be paid for being in this study?

You will be given up to \$30 in supermarket gift cards. You will get a \$10 gift card at the end of each session.

## Will being in this study cost you any money?

Being in this study will not cost you any money.

## What if you are hurt in this study?

If you are hurt as a result of being in this study, there are no plans to pay you for medical expenses, lost wages, disability, or discomfort. The charges for any medical treatment you receive will be billed to your insurance. You will be responsible for any amount your insurance does not cover. You do not give up any legal rights, such as seeking compensation for injury, by signing this form.

# What happens if you leave the study early?

You can change your mind about being in the study any time. You can agree to be in the study now and change your mind later. If you decide to stop being in the study, we will ask you to inform us immediately by calling or emailing the study team listed this form.

# How will your personal information be shared?

The UVA researchers are asking for your permission to gather, use and share information about you for this study. If you decide not to give your permission, you cannot be in this study, but you can continue to receive regular medical care at UVA.

# If you sign this form, we may collect any or all of the following information about you:

- o Personal information such as name and date of birth
- o Information collected about you from the questionnaires you complete.

UVA Study Tracking: HSR210100

Version Date: 03-22-21 Page Number: 4 of 7

#### Who will see your private information?

- The researchers to make sure they can conduct the study the right way, observe the effects of the study and understand its results
- o People or groups that oversee the study to make sure it is done correctly
- The sponsor(s) of this study, and the people or groups it hires to help perform or review this research
- o If you tell us that someone is hurting you, or that you might hurt yourself or someone else, the law may require us to let people in authority know so they can protect you and others.

Information about you may be given to other researchers outside of the University of Virginia after all identifiers such as name have been removed.

Some of the people outside of UVa who will see your information may not have to follow the same privacy laws that we follow. They may release your information to others, and it may no longer be protected by those laws.

The information collected from you might be published in a journal. This would be done in a way that protects your privacy. No one will be able to find out from the article that you were in the study.

Information obtained from you during this study will not be used in future research.

# What if you sign the form but then decide you don't want your private information shared?

You can change your mind at any time. Your permission does not end unless you cancel it. To cancel it, please send a letter to the researchers listed on this form or complete the "Leaving the Study Early" part of this form and return it to the researchers. Then you will no longer be in the study. The researchers will still use information about you that was collected before you ended your participation.

# Please contact the Principal Investigator listed earlier in this form to:

- Obtain more information about the study
- Ask a question about the study procedures or treatments
- Report an illness, injury, or other problem (you may also need to tell your regular doctors)
- Leave the study before it is finished
- Express a concern about the study

UVA Study Tracking: HSR210100

Version Date: 03-22-21 Page Number: 5 of 7

#### What if you have a concern about this study?

You may also report a concern about this study or ask questions about your rights as a research subject by contacting the Institutional Review Board listed below.

University of Virginia Institutional Review Board for Health Sciences Research PO Box 800483, Charlottesville, Virginia 22908, Telephone: 434-924-9634

When you call or write about a concern, please give as much information as you can. Include the name of the study leader, the IRB-HSR Number (at the top of this form), and details about the problem. This will help officials look into your concern. When reporting a concern, you do not have to give your name.

## **Signatures**

#### What does your signature mean?

Before you sign this form, please ask questions about any part of this study that is not clear to you. Your signature below means that you have received this information and all your

| PARTICIPANT | PARTICIPANT | <br>DATE |
|---|---|---|
| (SIGNATURE) | (PRINT) | |
| To be completed by participant | if 18 years of age or older. | |
| Person Obtaining Consent | | |
| Person Obtaining Consent By signing below you confirm the allowed them time to read the coall their questions. | • • | • |
| By signing below you confirm the allowed them time to read the co | • • | • |

UVA Study Tracking: HSR210100

Version Date: 03-22-21 Page Number: 6 of 7

# Leaving the Study Farly

| | Leaving the Study Lan | <u>Y</u> |
|---|---|---|
| Signatures should be obtained | ed in this section if the subject deci | des to leave the study early. |
| • | the study leader will keep the data help determine the results of the s | , . |
| | consent for this study. No addition p information from my medical red | • |
| Signature From Adult | | |
| PARTICIPANT (SIGNATURE) | PARTICIPANT (PRINT) | DATE |
| To be completed by particip | oant if 18 years of age or older. | |
| <b>Person Obtaining Signature</b> | | |
| By signing below you confirm | n that you have fully explained the | e implications of withdrawing |
| | t and have answered all their ques | |
| PERSON OBTAINING | PERSON OBTAINING | DATE |
| SIGNATURE | SIGNATURE | |
| (SIGNATURE) | (PRINT) | |

UVA Study Tracking: HSR210100 Version Date: 03-22-21 Page Number: 7 of 7